CLINICAL TRIAL: NCT06023732
Title: Behavioral Activation and Emotion-focused Interventions in the Treatment of Depression, A Single-case Study
Brief Title: Behavioral Activation and Emotion-focused Interventions in the Treatment of Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERDEP
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The research question will be investigated using a multiple baseline single-case A-B design. A will be the baseline phase, varying between 7 and 14 days, assessing the pattern of depression, behavioral activation and difficulties in emotion regulation before the intervention. Phase B comprise behavioral activation and emotion focused interventions as the independent variable and makes it possible to evaluate the effect of treatment on the dependent variable depressive symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Baseline 7 days (Experimental): Behavioral activation and emotion-focused interventions Baseline randomized length 7-14 days
  Interventions: Behavioral: Behavioral activation and emotion-focused interventions
- Baseline 8 days (Experimental): Behavioral activation and emotion-focused interventions Baseline randomized length 7-14 days
  Interventions: Behavioral: Behavioral activation and emotion-focused interventions
- Baseline 9 days (Experimental): Behavioral activation and emotion-focused interventions Baseline randomized length 7-14 days
  Interventions: Behavioral: Behavioral activation and emotion-focused interventions
- Baseline 10 days (Experimental): Behavioral activation and emotion-focused interventions Baseline randomized length 7-14 days
  Interventions: Behavioral: Behavioral activation and emotion-focused interventions
- Baseline 11 days (Experimental): Behavioral activation and emotion-focused interventions Baseline randomized length 7-14 days
  Interventions: Behavioral: Behavioral activation and emotion-focused interventions
- Baseline 12 days (Experimental): Behavioral activation and emotion-focused interventions Baseline randomized length 7-14 days
  Interventions: Behavioral: Behavioral activation and emotion-focused interventions
- Baseline 13 days (Experimental): Behavioral activation and emotion-focused interventions Baseline randomized length 7-14 days
  Interventions: Behavioral: Behavioral activation and emotion-focused interventions
- Baseline 14 days (Experimental): Behavioral activation and emotion-focused interventions Baseline randomized length 7-14 days
  Interventions: Behavioral: Behavioral activation and emotion-focused interventions

INTERVENTIONS:
Behavioral: Behavioral activation and emotion-focused interventions — Behavioral activation with emotion-focused interventions comprises two consecutive phases. In the first phase, treatment focus is behavioral activation in line with Brief behavioral activation treatment for depression - revised (BATD-R; 11) During the second phase, treatment focus shifts to address participants' emotions. Difficulties in understanding, tolerating, and labeling emotions is addressed by observing and describing emotions (12). Under the guidance of the therapist, participants are instructed to explore emotions normally avoided or ruminated on. This is conceptualized as a form of exposure to aversive emotions, thoughts and memories, to initiate emotional processing (13).

SUMMARY:
The study is a single-case intervention study, evaluating effects of the treatment Behavioral activation and emotion-focused interventions for depression.

Research question and hypothesis

1. What is the effect of behavioural activation and emotion-focused interventions on patients' ratings of depressive symptoms, behavioural activation and emotion regulation difficulties?
2. What is the effect of behavioural activation and emotion-focused interventions on patients' overall psychiatric state, with regards to ratings of anxiety, quality of life, level of functioning?
3. How does patient ratings of behavioural activation and emotion regulation difficulties and skills change during the course of treatment, in relation to treatment/session content?

DETAILED DESCRIPTION:
Procedure The study will be carried out by the authors or experienced clinicians (master level students at the Psychotherapy program at the Karolinska Institute), recruiting and treating patients with recurring depression at a primary care unit in the Stockholm region. 7 patients will be treated during 15 weeks. The treatment will be carried out in a blended format with an internet-based treatment supported with therapist face-to-face sessions. The initial behavioural activation phase lasts up to 6 weeks followed by additional emotion focused interventions. The treatment is initiated by a therapist session, thereafter therapist sessions are planned approximately every 3rd week.

To be included in the study participants must meet diagnostic criteria for depression as their primary problem according to DSM-5 (Diagnostic and Statistical Manual), have basic reading and writing skills in Swedish, and not express acute suicidal ideation. Patients with concurrent co-morbid psychiatric problems are eligible for inclusion unless another psychiatric diagnosis is assessed as primary to depression. Patients will be recruited from the regular flow of patients who seek treatment for psychological problems in the selected clinic. If interested they will be contacted by the study therapists and screened and assessed for eligibility after signing an informed consent.

Participants meeting inclusion criteria and not exclusion criteria will be offered participation in the study, and randomized to one of the 7 baseline lengths.

Methodology/approach/data analysis The research question will be investigated using a multiple baseline single-case A-B design. A will be the baseline phase, varying between 7 and 14 days, assessing the pattern of depression, behavioral activation and difficulties in emotion regulation before the intervention. Phase B comprise behavioral activation and emotion focused interventions as the independent variable and makes it possible to evaluate the effect of treatment on the dependent variable depressive symptoms. The B-phase will last 15 weeks and include the full internet-based treatment supported with 5-10 face-to-face therapist sessions .

Single-case experimental design (SCED) is particularly useful when evaluating a novel treatment in a clinical context as it produces reliable results even with a small sample size. Also, it is particularly helpful for studying the details of how the intervention works for each individual patient, through detailed and repeated measures of several dependent variables and processes. It is recommended that the effect of the intervention is assessed in at least 3 individuals (1), however, we will recruit at least 7 participants to allow for higher statistical power and as a safety measure for drop out and missing data.

Primary treatment effects in terms of depression, behavioural activation and emotion regulation will be assessed daily from day of inclusion to end of follow-up, with brief versions of self-rated measures with good reliability and validity. Brief versions of the following scales will be used for the daily assessment; depressive symptoms PHQ-2 (2), difficulties in emotion regulation, and daily behavioural activation BADS (3). Longitudinal data will be analyzed with non-parametric statistical tests (1). Visual inspection will be used to analyse variability, trends and patterns of change in the daily assessments over the phases of treatment.

Kendal's Tau is a non-overlap statistical test that has been developed for analysing SCED time series data with adequate statistical power. It will be used to analyse statistical differences in the dependent variables between phases. Kendal's Tau will be complemented with Tau-U tests if there are statistical trends in the data-series. Statistical power is very difficult to calculate for this test but given the expected medium effect sizes of the interventions and the replication across five participants, the statistical power is assessed as adequate. Pre, post and follow-up data will be assessed at start of phase A, start of phase B, after phase B and at follow up 3 months post treatment. The measures used will be PHQ-9 (4) for depression, GAD-7 (5) for anxiety symptoms, WSAS (6) for disability and ISI (7) for symptoms of insomnia. To measure if the treatment affects emotion regulation, self-ratings of DERS 16 (8) will be used. Post treatment the CSQ-8 (9) will be used to assess treatment satisfaction and NEQ (10) to asses negative effects.

ELIGIBILITY:
Inclusion Criteria:

* meet diagnostic criteria for depression as their primary problem according to DSM-5
* have basic reading and writing skills in Swedish
* not express acute suicidal ideation

Exclusion Criteria:

* concurrent comorbid psychiatric problems assessed as primary to depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2025-10-07 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-2 (PHQ-2) | Change from baseline (pre intervention start) to post intervention (15 weeks post intervention start)
  The PHQ-2 is a brief self-rating scale for screening major depression according to DSMIV and measuring current symptom level of depression. Min 0 max 6. Higher scores indicating more symptoms. The items correspond to the core criteria for depression in the DSM-IV.
  The scale can be used as screening for the criteria for a depressive syndrome may be present according to DSM-IV.
  You can also use the sum score as a measure of the current level of symptoms to assess the depth of depression and follow a course over time. The scale steps are scored from 0 to 3 and summed.
2 item Behavioral Activation for Depression Scale (BADS) | Change from baseline (pre intervention start) to post intervention (15 weeks post intervention start)
  The scale is designed to be administered weekly to measure changes over the course of Behavioral Activation for depression. The 2 most central items concerning rumination and behavioral activation are chosen and rated 0-6 from Not at all to Completely, where higher scores indicate more sufficient behavioral activation (less depressed behavior). Total score ranges from 0-12.
Emotion Regulation | Change from baseline (pre intervention start) to post intervention (15 weeks post intervention start)
  2 items regarding self rated emotion regulation. Items: Today I have been able to understand my emotions and needs, Today I have been able to accept my emotions and needs are rated from 1-5 where 1= Almost never and 5= Almost always. Total score ranges from 2-10 where higher scores indicate more sufficient emotion regulation.

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale, Brief Version (DERS-16) | Change from pre intervention to post intervention (15 weeks post intervention start)
  Self rated difficulties in emotion regulation. The sum ranges from 16 to 80, where higher levels indicate greater difficulty in emotion regulation.
Difficulties in Emotion Regulation Scale, Brief Version (DERS-16) | Change from pre intervention to post Behavioral activation phase (5 weeks post intervention start)
  Self rated difficulties in emotion regulation. The sum ranges from 16 to 80, where higher levels indicate greater difficulty in emotion regulation.
Difficulties in Emotion Regulation Scale, Brief Version (DERS-16) | Change from pre intervention to follow up 6 months post intervention start
  Self rated difficulties in emotion regulation. The sum ranges from 16 to 80, where higher levels indicate greater difficulty in emotion regulation.
Difficulties in Emotion Regulation Scale, Brief Version (DERS-16) | Change from pre intervention to follow up 12 months post intervention start
  Self rated difficulties in emotion regulation. The sum ranges from 16 to 80, where higher levels indicate greater difficulty in emotion regulation.
Patient Health Questionnaire (PHQ-9) | Change from pre intervention to post intervention (15 weeks post intervention start)
  The PHQ-9 is a brief self-rating scale for screening major depression according to DSMIV and measuring current symptom level of depression. Min 0 max 27. Higher scores indicating more symptoms. The first nine items in the PHQ-9 correspond to the nine criteria for depression in the DSM-IV. The tenth item is a simple function scale.
  The scale can be used as screening for the criteria for a depressive syndrome may be present according to DSM-IV.
  You can also use the sum score as a measure of the current level of symptoms to assess the depth of depression and follow a course over time. The scale steps for the first 9 items are scored from 0 to 3 and summed.
Patient Health Questionnaire (PHQ-9) | Change from pre intervention to post Behavioral activation phase (5 weeks post intervention start)
  The PHQ-9 is a brief self-rating scale for screening major depression according to DSMIV and measuring current symptom level of depression. Min 0 max 27. Higher scores indicating more symptoms. The first nine items in the PHQ-9 correspond to the nine criteria for depression in the DSM-IV. The tenth item is a simple function scale.
  The scale can be used as screening for the criteria for a depressive syndrome may be present according to DSM-IV.
  You can also use the sum score as a measure of the current level of symptoms to assess the depth of depression and follow a course over time. The scale steps for the first 9 items are scored from 0 to 3 and summed.
Patient Health Questionnaire (PHQ-9) | Change from pre intervention to post intervention follow up 6 months post intervention start
  The PHQ-9 is a brief self-rating scale for screening major depression according to DSMIV and measuring current symptom level of depression. Min 0 max 27. Higher scores indicating more symptoms. The first nine items in the PHQ-9 correspond to the nine criteria for depression in the DSM-IV. The tenth item is a simple function scale.
  The scale can be used as screening for the criteria for a depressive syndrome may be present according to DSM-IV.
  You can also use the sum score as a measure of the current level of symptoms to assess the depth of depression and follow a course over time. The scale steps for the first 9 items are scored from 0 to 3 and summed.
Patient Health Questionnaire (PHQ-9) | Change from pre intervention to follow up 12 months post intervention start
  The PHQ-9 is a brief self-rating scale for screening major depression according to DSMIV and measuring current symptom level of depression. Min 0 max 27. Higher scores indicating more symptoms. The first nine items in the PHQ-9 correspond to the nine criteria for depression in the DSM-IV. The tenth item is a simple function scale.
  The scale can be used as screening for the criteria for a depressive syndrome may be present according to DSM-IV.
  You can also use the sum score as a measure of the current level of symptoms to assess the depth of depression and follow a course over time. The scale steps for the first 9 items are scored from 0 to 3 and summed.
Behavioral Activation for Depression Scale (BADS) short version 9 items | Change from pre intervention to post intervention (15 weeks post intervention start)
  The questionnaire is designed to measure changes in avoidance and activation over the course of Behavioral Activation for depression. Items are rated from Not at all to Completely, where higher scores indicate more sufficient behavioral activation (less depressed behavior). Total score ranges from 0-54.
Behavioral Activation for Depression Scale (BADS) short version 9 items | Change from pre intervention to post Behavioral activation phase (5 weeks post intervention start)
  The questionnaire is designed to measure changes in avoidance and activation over the course of Behavioral Activation for depression. Items are rated from Not at all to Completely, where higher scores indicate more sufficient behavioral activation (less depressed behavior). Total score ranges from 0-54.
Behavioral Activation for Depression Scale (BADS) short version 9 items | Change from pre intervention to follow up 6 months post intervention start
  The questionnaire is designed to measure changes in avoidance and activation over the course of Behavioral Activation for depression. Items are rated from Not at all to Completely, where higher scores indicate more sufficient behavioral activation (less depressed behavior). Total score ranges from 0-54.
Behavioral Activation for Depression Scale (BADS) short version 9 items | Change from pre intervention to follow up 12 months post intervention start
  The questionnaire is designed to measure changes in avoidance and activation over the course of Behavioral Activation for depression. Items are rated from Not at all to Completely, where higher scores indicate more sufficient behavioral activation (less depressed behavior). Total score ranges from 0-54.
Generalized Anxiety Disorder 7-item scale (GAD-7) | Change from pre intervention to post intervention (15 weeks post intervention start)
  The GAD-7 is an instrument developed to help people who have anxiety symptoms that can be described as GAD. The test is only indicative and can never replace a doctor's visit and accurate diagnostics. The questions can be a help for the customer to identify any problems together with their doctor. If the client is already undergoing treatment for GAD, it may also be valuable to do a self-assessment from time to time to evaluate the effect of the treatment. A good opportunity can be in connection with and before a return visit to a doctor or psychologist or alternatively in connection with the renewal of a prescription. The customer can print out and take the test result to their doctor. The seven questions are scored from 0 (Not at all) to 3 (Daily) and summed. The total score is thus within the range 0-21.
Generalized Anxiety Disorder 7-item scale (GAD-7) | Change from pre intervention to post Behavioral activation phase (5 weeks post intervention start)
  The GAD-7 is an instrument developed to help people who have anxiety symptoms that can be described as GAD. The test is only indicative and can never replace a doctor's visit and accurate diagnostics. The questions can be a help for the customer to identify any problems together with their doctor. If the client is already undergoing treatment for GAD, it may also be valuable to do a self-assessment from time to time to evaluate the effect of the treatment. A good opportunity can be in connection with and before a return visit to a doctor or psychologist or alternatively in connection with the renewal of a prescription. The customer can print out and take the test result to their doctor. The seven questions are scored from 0 (Not at all) to 3 (Daily) and summed. The total score is thus within the range 0-21.
Generalized Anxiety Disorder 7-item scale (GAD-7) | Change from pre intervention to follow up 6 months post intervention start
  The GAD-7 is an instrument developed to help people who have anxiety symptoms that can be described as GAD. The test is only indicative and can never replace a doctor's visit and accurate diagnostics. The questions can be a help for the customer to identify any problems together with their doctor. If the client is already undergoing treatment for GAD, it may also be valuable to do a self-assessment from time to time to evaluate the effect of the treatment. A good opportunity can be in connection with and before a return visit to a doctor or psychologist or alternatively in connection with the renewal of a prescription. The customer can print out and take the test result to their doctor. The seven questions are scored from 0 (Not at all) to 3 (Daily) and summed. The total score is thus within the range 0-21.
Generalized Anxiety Disorder 7-item scale (GAD-7) | Change from pre intervention to follow up 12 months post intervention start
  The GAD-7 is an instrument developed to help people who have anxiety symptoms that can be described as GAD. The test is only indicative and can never replace a doctor's visit and accurate diagnostics. The questions can be a help for the customer to identify any problems together with their doctor. If the client is already undergoing treatment for GAD, it may also be valuable to do a self-assessment from time to time to evaluate the effect of the treatment. A good opportunity can be in connection with and before a return visit to a doctor or psychologist or alternatively in connection with the renewal of a prescription. The customer can print out and take the test result to their doctor. The seven questions are scored from 0 (Not at all) to 3 (Daily) and summed. The total score is thus within the range 0-21.
Insomnia Severity Index (ISI) | Change from pre intervention to post intervention (15 weeks post intervention start)
  A self-report questionnaire intended to measure insomnia. The purpose of the form is to quickly obtain a measure of the severity of sleep problems. The scale consists of 7 questions that evaluate falling asleep, sleep during the night, early awakening, the feeling of being rested, how sleep problems affect daily life and how the sleep pattern worries the individual. For each question, the participants must take a position on how they have experienced their sleeping habits in the past two weeks and then indicate the answers on a five-point Likert scale from 0 to 4, where 0 stands for "not at all" and 4 stands for "very much". The points are then added up. The total can be from 0 to 28 points. High scores indicate more severe sleep problems.
Insomnia Severity Index (ISI) | Change from pre intervention to post Behavioral activation phase (5 weeks post intervention start)
  A self-report questionnaire intended to measure insomnia. The purpose of the form is to quickly obtain a measure of the severity of sleep problems. The scale consists of 7 questions that evaluate falling asleep, sleep during the night, early awakening, the feeling of being rested, how sleep problems affect daily life and how the sleep pattern worries the individual. For each question, the participants must take a position on how they have experienced their sleeping habits in the past two weeks and then indicate the answers on a five-point Likert scale from 0 to 4, where 0 stands for "not at all" and 4 stands for "very much". The points are then added up. The total can be from 0 to 28 points. High scores indicate more severe sleep problems.
Insomnia Severity Index (ISI) | Change from pre intervention to follow up 6 months post intervention start
  A self-report questionnaire intended to measure insomnia. The purpose of the form is to quickly obtain a measure of the severity of sleep problems. The scale consists of 7 questions that evaluate falling asleep, sleep during the night, early awakening, the feeling of being rested, how sleep problems affect daily life and how the sleep pattern worries the individual. For each question, the participants must take a position on how they have experienced their sleeping habits in the past two weeks and then indicate the answers on a five-point Likert scale from 0 to 4, where 0 stands for "not at all" and 4 stands for "very much". The points are then added up. The total can be from 0 to 28 points. High scores indicate more severe sleep problems.
Insomnia Severity Index (ISI) | Change from pre intervention to follow up 12 months post intervention start
  A self-report questionnaire intended to measure insomnia. The purpose of the form is to quickly obtain a measure of the severity of sleep problems. The scale consists of 7 questions that evaluate falling asleep, sleep during the night, early awakening, the feeling of being rested, how sleep problems affect daily life and how the sleep pattern worries the individual. For each question, the participants must take a position on how they have experienced their sleeping habits in the past two weeks and then indicate the answers on a five-point Likert scale from 0 to 4, where 0 stands for "not at all" and 4 stands for "very much". The points are then added up. The total can be from 0 to 28 points. High scores indicate more severe sleep problems.
The Work and Social Adjustment Scale (WSAS) | Change from pre intervention to post intervention (15 weeks post intervention start)
  The WSAS is a simple, reliable and valid measure of impaired functioning. It is a sensitive and useful outcome measure offering the potential for readily interpretable comparisons across studies and disorders. The maximum score of the WSAS is 40, lower scores are better. The 5 items are scored 0-8 ranging from Not at-all-Slightly-Definitely-Markedly-Very-severely
The Work and Social Adjustment Scale (WSAS) | Change from pre intervention to post post Behavioral activation phase (5 weeks post intervention start)
  The WSAS is a simple, reliable and valid measure of impaired functioning. It is a sensitive and useful outcome measure offering the potential for readily interpretable comparisons across studies and disorders. The maximum score of the WSAS is 40, lower scores are better. The 5 items are scored 0-8 ranging from Not at-all-Slightly-Definitely-Markedly-Very-severely
The Work and Social Adjustment Scale (WSAS) | Change from pre intervention to follow up 6 months post intervention start
  The WSAS is a simple, reliable and valid measure of impaired functioning. It is a sensitive and useful outcome measure offering the potential for readily interpretable comparisons across studies and disorders. The maximum score of the WSAS is 40, lower scores are better. The 5 items are scored 0-8 ranging from Not at-all-Slightly-Definitely-Markedly-Very-severely
The Work and Social Adjustment Scale (WSAS) | Change from pre intervention to follow up 12 months post intervention start
  The WSAS is a simple, reliable and valid measure of impaired functioning. It is a sensitive and useful outcome measure offering the potential for readily interpretable comparisons across studies and disorders. The maximum score of the WSAS is 40, lower scores are better. The 5 items are scored 0-8 ranging from Not at-all-Slightly-Definitely-Markedly-Very-severely
Client Satisfaction Questionnaire (CSQ-8) | Immediately post intervention
  Self rated questionnaire to rate satisfaction with treatment. 8 items rated from 1-4 and summarized. Lower scores indicating less satisfaction. Scale ranging from 0-32
Negative Effects Questionnaire (NEQ) | Immediately post intervention
  self-rating form to measure negative effects of psychological treatment The NEQ consists of 20 statements that are answered on a 0-4 Likert scale. Furthermore, there is an open question to try to capture such negative effects that are not included in the self-report form, but which may be of theoretical or clinical relevance. In addition, the respondent is asked to answer whether the negative effects experienced were due to the treatment they underwent or other circumstances. The scale ranges from 0-80, higher scores indicate more negative effects. However the scale is more descriptive than designed to calculate negative effects

CONTACTS AND LOCATIONS:
Locations (1):
- Liljeholmens primary care centre, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dugard P, File, P., Todman, J. Singel-case and Small-n experimental designs. New york: Routledge; 2001.
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Kanter JW, Mulick PS, Busch AM, Berlin KS, Martell CR. The Behavioral Activation for Depression Scale (BADS): Psychometric Properties and Factor Structure. Journal of Psychopathology and Behavioral Assessment. 2006;29(3):191.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Bjureberg J, Ljotsson B, Tull MT, Hedman E, Sahlin H, Lundh LG, Bjarehed J, DiLillo D, Messman-Moore T, Gumpert CH, Gratz KL. Development and Validation of a Brief Version of the Difficulties in Emotion Regulation Scale: The DERS-16. J Psychopathol Behav Assess. 2016 Jun;38(2):284-296. doi: 10.1007/s10862-015-9514-x. Epub 2015 Sep 14. PMID 27239096
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] Rozental A, Kottorp A, Forsstrom D, Mansson K, Boettcher J, Andersson G, Furmark T, Carlbring P. The Negative Effects Questionnaire: psychometric properties of an instrument for assessing negative effects in psychological treatments. Behav Cogn Psychother. 2019 Sep;47(5):559-572. doi: 10.1017/S1352465819000018. Epub 2019 Mar 15. PMID 30871650
- [Background] Lejuez CW, Hopko DR, Acierno R, Daughters SB, Pagoto SL. Ten year revision of the brief behavioral activation treatment for depression: revised treatment manual. Behav Modif. 2011 Mar;35(2):111-61. doi: 10.1177/0145445510390929. PMID 21324944
- [Background] Linehan MM. Cognitive Behavioral Treatment of Borderline Personality Disorder. New York: Guilford Press; 1993.
- [Background] Greenberg, Leslie S. and Goldman, Rhonda N. Clinical Handbook of Emotion-Focused Therapy. American Psychological Association. (2018).